CLINICAL TRIAL: NCT03656289
Title: Antepartum Etonogestrel Contraceptive Implant Insertion at Term: an Acceptability and Pharmacokinetic Pilot Study
Brief Title: Antepartum Etonogestrel Contraceptive Implant Insertion at Term
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: IND approval from FDA was rejected and IRB approval was never granted.
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 18-0197
Record Dates: First submitted 2018-08-23; First posted 2018-09-04 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Contraception
Keywords: Contraception; Etonogestrel implant
MeSH Terms: interventions — etonogestrel; Drug Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Etonogestrel Contraceptive (Experimental): Etonogestrel contraceptive implant; consists of a single, radiopaque, rod-shaped implant, containing 68 mg etonogestrel, pre-loaded in the needle of a disposable applicator. The implant must be removed no later than by the end of the third year.
  Interventions: Drug: Etonogestrel 68Mg Implant

INTERVENTIONS:
Drug: Etonogestrel 68Mg Implant — Participants will have an etonogestral contraceptive implant (NEXPLANON) placed sub-dermally just under the skin at the inner side of the non-dominant upper arm.
  Other Names: NEXPLANON

SUMMARY:
Short-interval pregnancy (SIP) or rapid, repeat pregnancy is defined as a pregnancy within one year of prior delivery. These pregnancies are often unintended and are associated with adverse risks. Low contraceptive initiation during the postpartum period is a contributing factor to SIP. This study will be the first to investigate the initiation of a highly-effective, immediately active contraceptive device during the antepartum period. The antepartum period serves as an ideal time for postpartum contraception counseling, due to patients' active involvement with the healthcare system. The pharmacokinetic analysis proposed in this study will be the first to investigate whether and to what extent ENG hormone crosses the placenta. This data will enrich understanding of the pharmacology of exogenous progestins administered during pregnancy and provide information that can be incorporated into future patient counseling regarding the risks of fetal exposure with exogenous progestin use.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women (ages 18-34 years) ≥37 weeks gestational age who are interested in using an ENG contraceptive implant for their postpartum birth control method.
* Women with a history of at least one uncomplicated vaginal delivery at term who have received routine prenatal care (at least five visits) including an anatomy ultrasound with confirmed dating.

Exclusion Criteria:

* Women outside the gestational age outlined above.
* Women who are seen outside of the enrolling clinics.
* Women 35 years and older at the time of anticipated delivery, as these women meet the clinical definition of advanced maternal age which has been associated with increased adverse events in pregnancy.
* Women with any condition that necessitates a medically indicated delivery (e.g. diabetes mellitus, any hypertensive disorder), multiple gestations, fetal anomalies, Class III obesity (body mass index >40), concurrent use of either an injectable or vaginal progestin, and any concerns related to ENG implant use based on the US Medical Eligibility Criteria for Contraceptive Use (defined as a class 3 or 4 recommendation).

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — We are only enrolling women in this study as we are studying the acceptability of a contraceptive device during pregnancy and so this study is not appropriate for men.
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Maternal and cord blood serum etonogestrel concentration | Delivery
  Maternal and cord blood serum etonogestrel concentratration

SECONDARY OUTCOMES:
Gestational age at time of delivery | Delivery
  Gestational age at time of delivery
Onset of lactogenesis | 5-10 days postpartum (Follow Up Visit 1)
  Stage II of lactation
Questionnaire: Continuation of contraceptive implant use | 3 months postpartum (Follow Up Visit 2)
  Assess continuation of the contraceptive implant
Questionnaire: Satisfaction with contraceptive implant | 3 months postpartum (Follow Up Visit 2)
  Assess satisfaction with the contraceptive implant
Questionnaire: Continuation of contraceptive implant use | 6 months postpartum (Follow Up Visit 3)
  Assess continuation of the contraceptive implant
Questionnaire: Satisfaction with contraceptive implant | 6 months postpartum (Follow Up Visit 3)
  Assess satisfaction with the contraceptive implant

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Lazorwitz, MD, Principal Investigator — University of Colorado - Denver Anschutz
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No